CLINICAL TRIAL: NCT07164521
Title: The Effect of Music Played During the Postoperative Period on Pain and Anxiety Levels in Women Who Underwent Cesarean Delivery: A Randomized Controlled Trial
Brief Title: The Effect of Music Postoperative Period
Acronym: EMPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bihter Akın, Assoc. Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/647
Record Dates: First submitted 2025-08-31; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section; Dehiscence; Postoperative Pain
Keywords: Postoperative Pain; Cesarean Section; Anxiety
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group, which received music listening, or the control group, with no intervention, in a parallel assignment model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Music Listening (Experimental): Women in the intervention group listened to relaxing classical instrumental music (e.g., works by Mozart, Vivaldi, and Debussy) for 15 minutes every hour, starting at the 24th postpartum hour until the 48th hour.
  Interventions: Behavioral: Music Listening (Relaxing Classical Music)
- No Intervention - Control (No Intervention): Women in the control group received routine postpartum care without any additional intervention.

INTERVENTIONS:
Behavioral: Music Listening (Relaxing Classical Music) — Participants listened to a standardized playlist of relaxing classical instrumental music (e.g., Mozart, Vivaldi, Debussy) for 15 minutes every hour, beginning at the 24th postpartum hour until the 48th hour. The intervention aimed to reduce postpartum anxiety and pain perception.
  Other Names: Experimental - Music Listening
  Arms: Experimental - Music Listening

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of music listening on anxiety and pain among women following cesarean delivery. A total of 110 women who had undergone cesarean section were included. Beginning at the 24th postpartum hour, participants in the intervention group listened to relaxing classical music for 15 minutes every hour, while no intervention was applied to the control group. The study was designed to determine whether music listening could influence postpartum anxiety and perceived pain.

DETAILED DESCRIPTION:
Postpartum women undergoing cesarean section often experience significant levels of anxiety and pain, which can negatively affect recovery and maternal-infant bonding. In addition to pharmacological methods, non-pharmacological strategies such as music listening may play an important role in supporting women during this period. In this study, 110 women who had undergone cesarean delivery were randomly assigned to intervention and control groups. Starting at the 24th postpartum hour until the 48th hour, women in the intervention group listened to relaxing classical instrumental music (e.g., works by Mozart, Vivaldi, and Debussy) for 15 minutes every hour. The control group received no intervention. Participants' demographic and clinical characteristics were collected using the Descriptive Characteristics Form, while postpartum anxiety and pain perception were assessed with the Postpartum-Specific Anxiety Scale (PSAS) and Pain Catastrophizing Scale (PCS). The primary outcome was anxiety, and the secondary outcome was pain perception. The study sought to assess whether a music-based, culturally appropriate, non-pharmacological intervention could be an effective component of routine postpartum care following cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older

Primiparous (first-time mothers)

Underwent cesarean section under spinal anesthesia

Mentally healthy and able to communicate

No hearing impairments (able to hear the music intervention)

No chronic illnesses

No complications during labor for mother or newborn

Proficient in Turkish

Voluntarily agreed to participate and provided informed consent

Exclusion Criteria:

Multiparous women (previous childbirth experience)

Women who used non-routine analgesics beyond standard postpartum pain relievers

Presence of psychiatric disorders or severe mental illness

Medical complications during or after delivery for mother or infant

Hearing impairments preventing participation in music listening

Women unwilling or unable to comply with the intervention protocol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Postpartum Anxiety | 48th postpartum hour
  Measured using the Postpartum-Specific Anxiety Scale (PSAS) at the 48th postpartum hour. Higher scores indicate higher levels of anxiety.
Pain Catastrophizing | 48th postpartum hour
  Measured using the Pain Catastrophizing Scale (PCS) at the 48th postpartum hour. Higher scores indicate greater pain catastrophizing.

SECONDARY OUTCOMES:
Total Duration of Music Listening | Between the 24th and 48th postpartum hour
  Total number of minutes of music listened by participants in the intervention group across the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.

REFERENCES:
- [Derived] Akin B, Ozdemir S. The Effect of Music Played During the Postoperative Period on Pain and Anxiety Levels in Women Who Underwent Cesarean Delivery: A Randomized Controlled Trial. J Integr Complement Med. 2025 Oct 28. doi: 10.1177/27683605251389490. Online ahead of print. PMID 41182331